CLINICAL TRIAL: NCT07189910
Title: Efficacy and Safety of Glucocorticoids Combined With Recombinant Human Thrombopoietin (rhTPO) Sequential Eltrombopag Olamine for Severe Primary Immune Thrombocytopenia (ITP) in Adults
Brief Title: Sequential rhTPO and Eltrombopag Following Glucocorticoids for Severe Adult ITP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, MEI HENG, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITP-TPO+Eltro
Record Dates: First submitted 2025-08-12; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: immune thrombocytopenia (ITP); recombinant human thrombopoietin (rhTPO); Eltrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eltrombopag Group (Experimental): Participants who achieve a complete response (CR) or response (R) after HD-DXM combined with rhTPO treatment will be randomized in a 2:1 ratio into the eltrombopag group or the placebo group.
  Observation group: Participants will receive eltrombopag for oral suspension (EPAG-pfos) for ten weeks.
  Interventions: Drug: Eltrombopag
- Placebo group (Active Comparator): Participants who achieve a complete response (CR) or response (R) after HD-DXM combined with rhTPO treatment will be randomized in a 2:1 ratio into the eltrombopag group or the placebo group.
  Control group: Participants did not receive sequential EPAG-pfos treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Participants assigned to the observation group will be treated with eltrombopag oral suspension (EPAG-pfos).
  Other Names: EPAG-pfos
  Arms: Eltrombopag Group
Other: Placebo — Participants in the control group will receive a placebo at the same dose, instead of eltrombopag oral suspension (EPAG-pfos).
  Arms: Placebo group

SUMMARY:
To address the clinical need for improving early response rates, maintaining sustained responses, reducing relapse rates, and minimizing adverse events in the treatment of immune thrombocytopenia (ITP), the investigators developed a comprehensive in-hospital and post-discharge management strategy. In this study, hospitalized participants will receive a 14-day regimen of high-dose dexamethasone (HD-DXM) plus recombinant human thrombopoietin (rhTPO), followed by a 10-week course of oral eltrombopag olamine dry suspension after discharge. The investigators aim to evaluate the efficacy and safety of this sequential treatment strategy in adult ITP patients.

DETAILED DESCRIPTION:
To address the clinical need for improving early response rates, maintaining sustained responses, reducing relapse rates, and minimizing adverse events in the treatment of immune thrombocytopenia (ITP), the investigators developed a comprehensive in-hospital and post-discharge management strategy. This approach is based on the superior early response achieved with recombinant human thrombopoietin (rhTPO) combined with high-dose dexamethasone (HD-DXM), and the favorable efficacy of eltrombopag in maintaining long-term responses and reducing relapse. In this study, hospitalized participants will receive a 14-day regimen of HD-DXM plus rhTPO, followed by a 10-week course of oral eltrombopag olamine dry suspension after discharge. The investigators aim to evaluate the efficacy and safety of this sequential treatment strategy in adult ITP participants, with the goal of enhancing early response, sustaining remission, reducing relapse, and minimizing adverse effects. This study is expected to provide evidence-based support for optimizing ITP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 75 years, regardless of gender;
* ECOG performance status of 0-1;
* Diagnosis of primary ITP confirmed by bone marrow biopsy (valid within 3 months) and other relevant assessments; baseline platelet count (PLT) <20×10⁹/L within 48 hours prior to administration of study medication;
* Adequate function of major organs as defined below (based on the clinical laboratory reference ranges of the study center):
* Hematology: Absolute neutrophil count (ANC) ≥1.5×10⁹/L; no abnormalities unrelated to ITP, except a) PLT <20×10⁹/L at Day 1 or within 48 hours of Day 1 is allowed; b) Hemoglobin: If anemia is clearly due to ITP-related bleeding, hemoglobin lower than the lower limit of normal (LLN) may be permitted at investigator's discretion.
* Biochemistry: Total bilirubin (TBIL) ≤1.5×ULN; ALT, AST, ALP ≤3×ULN; serum creatinine ≤1.5×ULN and creatinine clearance ≥50 mL/min.
* Coagulation: Prothrombin time (PT) within ±3 seconds of normal range; activated partial thromboplastin time (APTT) ≤1.5×ULN unless on medications known to alter INR/APTT; no known history of coagulopathy other than ITP.
* Prior ITP rescue treatments (e.g., platelet transfusion, IVIG, immunomodulators, cyclophosphamide) must have ended or failed at least 2 weeks prior to enrollment (except corticosteroids); TPO-RAs or corticosteroids must be discontinued ≥14 days before study start.
* Patients on maintenance immunosuppressive therapy (e.g., corticosteroids, azathioprine, danazol, cyclosporine A, mycophenolate mofetil, or traditional Chinese platelet-raising medicine) must be on stable doses for at least 1 month prior to enrollment. Patients previously treated with anti-CD20 antibodies must have discontinued at least 6 months prior; splenectomy patients may enroll ≥6 months post-surgery.
* Female subjects of childbearing potential must have a negative serum pregnancy test within 24 hours prior to first dosing; all subjects agree to use effective contraception during the study and for 6 months after its completion.
* No known contraindications to corticosteroids, rhTPO, or eltrombopag and willing to undergo rhTPO followed by eltrombopag treatment.
* Willingness to participate and ability to provide written informed consent. For participants aged ≥12 years, both the subject and their legal guardian must sign the informed consent form.

Exclusion Criteria:

* Refractory ITP (failure to respond to first- and second-line TPO-RAs, anti-CD20 therapy, or splenectomy);
* Pregnant or lactating women;
* Evidence of secondary ITP (e.g., untreated Helicobacter pylori, leukemia, lymphoma, autoimmune diseases such as SLE, Hashimoto's thyroiditis), drug-induced thrombocytopenia (e.g., due to anticonvulsants, antibiotics, heparin), or multi-lineage autoimmune cytopenias (e.g., Evans syndrome);
* History or presence of any primary disease other than ITP that may cause thrombocytopenia (e.g., myelodysplastic syndrome, congenital bone marrow failure syndromes such as Fanconi anemia or dyskeratosis congenita, aplastic anemia), as judged by the investigator;
* History of intracranial hemorrhage or severe bleeding (>CTCAE Grade 3) of vital organs; symptomatic gastrointestinal bleeding (e.g., hematemesis, melena) within 6 months prior to screening (asymptomatic occult blood and hemorrhoids excluded);
* History of any arterial or venous thrombosis (e.g., stroke, TIA, MI, DVT, PE) within 6 months prior to enrollment and at least two of the following risk factors: hormone replacement therapy, oral contraceptives (including estrogens), smoking, diabetes, hypercholesterolemia, pharmacologically controlled hypertension, hereditary thrombophilia;
* Severe cardiovascular disease within 6 months prior to enrollment (e.g., NYHA Class III-IV), arrhythmias increasing thrombotic risk (e.g., atrial fibrillation), or history of coronary stenting, angioplasty, or bypass surgery;
* Concurrent serious or life-threatening malignancy;
* Use of drugs that significantly affect platelet function (e.g., aspirin, clopidogrel, NSAIDs) or anticoagulants for >3 days within 2 weeks before and during the study;
* Use of any herbal medicine or nutritional supplement within 1 week prior to study start, except for vitamins and minerals;
* Ongoing or uncontrolled serious infections (≥CTCAE Grade 2);
* Laboratory or clinical evidence of HIV infection, active hepatitis C, active hepatitis B, or previous history of these infections. Patients with positive HBsAg are excluded. Those with HBsAg-negative but HBcAb-positive must undergo HBV DNA testing; if positive, they are excluded;
* Any condition deemed by the investigator to make the subject unsuitable for participation, including but not limited to medical, social, or psychological factors affecting safety or study compliance.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained response rate (SRR) at 3 months of treatment. | 3 months of the study
  Sustained response rate (SRR) at 3 months of treatment.

SECONDARY OUTCOMES:
The proportions of patients achieving response (R); | 6 months of the study
  The proportions of patients achieving response (R);
Platelet count levels at 3 months after treatment | 3 months of the study
  Platelet count levels at 3 months after treatment
The proportions of patients achieving complete response (CR); | 6 months of the study
  The proportions of patients achieving complete response (CR);
The proportions of patients achieving and platelet counts ≥50×10⁹/L; | 6 months of the study
  The proportions of patients achieving and platelet counts ≥50×10⁹/L;
Sustained response rate (SRR) at 6 months; | 6 months of the study
  Sustained response rate (SRR) at 6 months;
Time to response (TTR); | 6 months of the study
  Time to response (TTR);
Time from treatment initiation to first achievement of PLT ≥100×10⁹/L; | 6 months of the study
  Time from treatment initiation to first achievement of PLT ≥100×10⁹/L;

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
It is not clear whether the data would involve patient privacy or whether patients would agree to the disclosure of the data.